CLINICAL TRIAL: NCT02052557
Title: The Effect of Exparel on Post Operative Pain and Narcotic Use After Colon Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Des Moines University (Other)
Collaborators: Mercy Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MMC2013-09
Record Dates: First submitted 2014-01-24; First posted 2014-02-03 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Post-operative Pain; Colon Cancer; Diverticulitis
Keywords: Exparel; liposomal bupivicaine; post operative pain control; local anesthetic after surgery; colorectal surgery; marcaine; long acting local anesthetic; pain medication use after surgery
MeSH Terms: conditions — Pain, Postoperative; Colonic Neoplasms; Diverticulitis | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): 30 milliliters (ml) of 0.5% marcaine with epinephrine
  Interventions: Drug: Bupivacaine
- Bupivacaine liposome suspension (Active Comparator): exparel 20ml, diluted with 10ml sterile saline for total of 30ml
  Interventions: Drug: Bupivacaine liposome suspension

INTERVENTIONS:
Drug: Bupivacaine — 30ml of bupivacaine were injecting into the subcutaneous tissue at the incision sites after surgery in the OR
  Other Names: Marcaine
  Arms: Bupivacaine
Drug: Bupivacaine liposome suspension — 30ml of Bupivacaine liposome injectable suspension were injecting into the subcutaneous tissue at the incision sites after surgery in the OR
  Other Names: Exparel; 72 hour Bupivacaine; Long acting Bupivacaine
  Arms: Bupivacaine liposome suspension

SUMMARY:
The purpose of the study is to evaluate the effect of Exparel on pain control and patient outcome after colon resection. The investigators will evaluate the clinical course of the patients who receive exparel as compared to the patients who do not receive exparel. Exparel is a 72 hour bupivacaine which is slowly released from lysosomes over the course of three days. A long acting local anesthetic should provide better pain control than conventional bupivacaine which has a 3.5 hour half-life.

DETAILED DESCRIPTION:
Patients who are undergoing elective colon resection with Dr. Kraemer and Dr. Raman will be offered participation in the study. This will include robotic, laparoscopic and open procedures.

In the pre-operative area prior to surgery, the surgical resident will inform the patient of the opportunity to participate in the research study. The resident will consent the patient at that time, if the patient chooses to participate, they will be randomized to an exparel or non-exparel group. The randomization will be done by having the resident pick an envelope that will state whether or not the patient is randomized to the exparel or non-exparel group, this will randomize to 50% in each group. The patient will not be notified of the type of local anesthetic they receive. The attending surgeon will also be blind to the type of local the pt will receive; only the resident and Operating Room (OR) staff will know what type of local anesthetic was given. Unfortunately the opaque color of the exparel precludes the physician injecting the local anesthetic from being blinded to the type of anesthetic given.

The patient will be taken to the operating room as usual, and the surgery will proceed as it normally would. At the end of the surgery the patient will receive either exparel or bupivacaine depending upon which the patient was randomized to. The attending surgeon will not be in the operating suite while the local anesthetic is being injected. 30 milliliters (mL) of either exparel or bupivacaine will be injected into the subcutaneous tissues at the end of surgery.

The patient will be taken to the post operative care unit (PACU), the medications for post-operative pain will be standardized between the two groups, a standard starting dose on the patient controlled analgesia (PCA) will be used, and will be adjusted as needed. The postoperative care will attempt to be standardized in regard to diet, discharge (dc) of foley, not using nasogastric (NG) tubes, however this will be based on the individual patient was what is best for their care. This data will then be analyzed to determine if exparel has a beneficial effect on surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Elective colon resection for both benign and malignant disease
* Laparoscopic, robotic and open techniques

Exclusion Criteria:

* emergent colon cases
* cases preformed by surgeons other than Dr. Raman or Dr. Kraemer
* pregnant patients
* patients currently breast feeding
* patients under the age of 18
* other patients unable to give informed consent
* bupivacaine use within 96 hours
* allergy to amide anesthetics
* prisoners
* caution will be used in patients with renal or hepatic failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Knudson, DO, Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Des Moines, Iowa, United States

REFERENCES:
- [Derived] Knudson RA, Dunlavy PW, Franko J, Raman SR, Kraemer SR. Effectiveness of Liposomal Bupivacaine in Colorectal Surgery: A Pragmatic Nonsponsored Prospective Randomized Double Blinded Trial in a Community Hospital. Dis Colon Rectum. 2016 Sep;59(9):862-9. doi: 10.1097/DCR.0000000000000648. PMID 27505115

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants] — Population: The study personnel have left the institution or are unreachable. efforts were made to contact the PI/study team members but were unsuccessful. Efforts were also made to get data from Mercy IRB and patient records staff. These staff did not have the information to find such data. Available data from the publication has been entered, but no other data is available and all efforts to locate the data have been exhausted.
Age, Continuous [Mean (Standard Deviation); unit: years] — The study personnel have left the institution or are unreachable. efforts were made to contact the PI/study team members but were unsuccessful. Efforts were also made to get data from Mercy IRB and patient records staff. These staff did not have the information to find such data. Available data from the publication has been entered, but no other data is available and all efforts to locate the data have been exhausted.
  years | 67 (2) | 67 (2) | 67 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: PCA (Patient Controlled Analgesia) Usage
Description: Will measure the amount of PCA use for the first 48 hours after surgery.
Time Frame: 48 hours post operatively
Population: The study personnel have left the institution or are unreachable. efforts were made to contact the PI/study team members but were unsuccessful. Efforts were also made to get data from Mercy IRB and patient records staff. These staff did not have the information to find such data. Available data from the publication has been entered, but no other data is available and all efforts to locate the data have been exhausted.
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Oral Pain Medications
Description: the amount of post operative oral narcotic is measured post op
Time Frame: 48 hours postoperatively
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Total IV (Intravenous) Narcotic Used
Description: the total amount of IV narcotic is measured that is given during post op period prior to discharge
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Total Oral Narcotic Used
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Length of Stay
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days
Measure: Number; unit: days
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 26 | 25
days | 4 | 6

6. Secondary Outcome: Return of Bowel Function
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days, and the timing of return of bowel function returning will be recorded
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Readmission
Time Frame: 30 days post operative readmission
Population: No one readmitted.
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

8. Secondary Outcome: Toradol Use
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine Liposome Suspension | Bupivacaine
Number analyzed (Participants) | 26 | 25
Participants | 1 | 0

9. Secondary Outcome: Ofirmev
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days, and the amount of ofirmev used during admission will be recorded
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Nausea Medication
Time Frame: The amount of nausea medicine used 48 hours post op was recorded
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Foley Catheter Removal
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days, the timing of foley catheter removal will be recorded
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Postoperative Pain
Description: The investigators will talk to the patient after surgery immediately post operatively Post Operative Day (POD) #3-5 and POD #13-15 and ask the patients to rate their pain on a scale of 1-10.
Time Frame: POD #3-5 and POD #13-15
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Post Operative Satisfaction
Description: The investigators will ask the patient to rate their satisfaction with pain control.
Time Frame: POD #3-5 and POD #13-15
Population: as for outcome 1
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Home Oral Narcotic Use
Description: The investigators will ask the patients how many of their narcotic pain pills they used after surgery up to the POD #13-15
Time Frame: POD #13-15
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine Liposome Suspension | Bupivacaine
Number analyzed (Participants) | 25 | 26
Participants | 2 | 5

15. Other Pre Specified Outcome: NG (Nasogastric) Placement
Description: We recorded if an NG was placed immediately post operatively
Time Frame: POD #0 if NG was placed
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The study personnel have left the institution or are unreachable. efforts were made to contact the PI/study team members but were unsuccessful. Efforts were also made to get data from Mercy IRB and patient records staff. These staff did not have the information to find such data. Available data from the publication has been entered, but no other data is available and all efforts to locate the data have been exhausted.
Description: The study personnel have left the institution or are unreachable. efforts were made to contact the PI/study team members but were unsuccessful. Efforts were also made to get data from Mercy IRB and patient records staff. These staff did not have the information to find such data. Available data from the publication has been entered, but no other data is available and all efforts to locate the data have been exhausted.
Arm/Group | Bupivacaine | Bupivacaine Liposome Suspension
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No